CLINICAL TRIAL: NCT00461721
Title: Pilot Trial to Elaborate a Cutaneous Antigen Neutralization Test in Patients Suffering From Rhinoconjunctivitis Due to Grass Pollen During Immunotherapy
Brief Title: Pilot Trial to Elaborate a Cutaneous Antigen Neutralization Test in Patients Suffering From Rhinoconjunctivitis
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Other Study IDs: ZU-AgNT-003
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

SUMMARY:
To find a test to elaborate a parameter for specific immunotherapy in allergic patients

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Signed informed consent
* SIT 2000/2001
* 10 patients with SIT with a good result- 10 patients with bad results

Exclusion criteria:

* Pregnancy and breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: x
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-01 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Department of Dermatology, Zurich, Switzerland